CLINICAL TRIAL: NCT03894670
Title: Evaluation of Methods for Measuring Gastrointestinal Transit and Food Reward in Healthy Individuals - The PRESET Study
Acronym: PRESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristine Færch (Other)
Collaborators: University of Copenhagen (Other); IMotions A/S (Industry); University of Leeds (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kristine Færch, Senior Researcher and Team Leader, PhD, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-18026293
Record Dates: First submitted 2019-03-12; First posted 2019-03-28 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Healthy Participants
Keywords: Gastric emptying; Gastrointestinal transit; Food reward; Food preferences
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: The study is a randomized cross-over study including 15 healthy normal-weight individuals. On two separate test days participants ingest the SmartPill™ in combination with a SmartBar™ (standard procedure, reference) or a standard mixed breakfast meal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmartBar™ (Active Comparator): The wireless capsule technology, SmartPill™, is usually ingested together with a SmartBar™ which is a snack bar with a nutrient composition that differs substantially from a normal western diet.
  Interventions: Other: SmartBar™
- Standard mixed breakfast meal (Experimental): The SmartPill™ is ingested together with a standard mixed breakfast meal and the outcomes of interest will be compared with the SmartBar™ condition (reference).
  Interventions: Other: Standard mixed breakfast meal

INTERVENTIONS:
Other: Standard mixed breakfast meal — The standard mixed breakfast meal consists of:
  150 g yoghurt, 20 g muesli; 50 g wheat bun; 22 g rye bread; 25 g cheese; 25 g marmalade; 8 g butter; Total energy content: 500 kcal Macronutrient composition: 34 E% fat, 17 E% protein, 49 E% carbohydrate
  Arms: Standard mixed breakfast meal
Other: SmartBar™ — SmarBar™ (Medtronic, North Haven, MA, USA). Weight: 72 g; Total energy content: 260 kcal Macronutrient composition: 7 E% fat, 19 E% protein, 74 E% carbohydrate.
  Arms: SmartBar™

SUMMARY:
The wireless motility capsule technology, SmartPill™, can be used to assess gastric emptying and gastrointestinal (GI) transit time. The SmartPill is usually ingested together with a SmartBar™ which is a snack bar with a nutrient composition that differs substantially from a normal western diet. The primary aim of the present study is to compare effects of a SmartBar™ and a standard mixed meal on gastric emptying and GI motility.

DETAILED DESCRIPTION:
Background: The wireless motility capsule technology, SmartPill™, can be used to assess GI transit time including gastric emptying and small and large bowel transit time based on measurements of pH, pressure and temperature. The SmartPill™ allows for GI motility measurements under free-living conditions without radiation. The SmartPill is usually ingested together with a SmartBar™ which is a snack bar with a nutrient composition that differs substantially from a normal western diet. GI motility in response to meals plays an important role in regulation of e.g. appetite and glucose metabolism. Changes in appetite and metabolism in response to interventions are often assessed using a meal test and GI motility is assessed at the research facilities. The use of SmartPill™ in combination with a meal test would allow for assessment of GI motility under subsequent free-living conditions and improve our understanding of the effects of interventions on the integrative relationship between food intake, GI motility and metabolism. Most of our daily decisions and actions affecting energy intake are driven by the non-conscious processes; however, appetite is often assessed from participants' self-report which is associated with limitations such as desire to report socially desirable answers. Little is known about the complex interrelationship between biological markers of appetite e.g. GI hormones and subjective and objective measures of food related behavior under fasting and fed conditions.

The PRESET study has the following objectives:

1. To compare effects of a SmartBar™ and a standard mixed breakfast meal on gastric emptying and GI transit time measured using the SmartPill™ in normal-weight individuals.
2. To compare effects of a SmartBar™ and a standard mixed breakfast meal on concentrations of metabolites and pancreatic and GI hormones, and subjective and objective measures of appetite, food reward and food related behavior assessed from biometric responses (facial expression, galvanic skin response and eye tracking) to visual food stimuli varying in fat content and taste during the computerized Leeds Food Preference Questionnaire (LFPQ) in normal-weight individuals.
3. To assess potential associations between gastric emptying and GI motility, biological markers of appetite and subjective appetite and objective measures of food related behavior from biometric responses to visual food stimuli during the LFPQ in the fasting state and in response to meals in normal-weight individuals.

Testing includes assessments in the fasting state and in response to consumption of the SmartBar™ and a standard mixed meal (4-hour meal tests and subsequent 6-days free-living assessment period) on two separate test days.

ELIGIBILITY:
Inclusion Criteria:

• Body mass index: 18.5 to 24.9 kg/m2

Exclusion Criteria:

* Unable to understand the informed consent and the study procedures;
* Self-reported history of an eating disorder in the past three years
* Self-reported weight change (>5 kg) within three months prior to inclusion
* HbA1c: ≥5.7 % (≥39 mmol/mol)
* Uncontrolled medical issues including but not limited to cardiovascular pulmonary, rheumatologic, hematologic, oncologic, infectious, GI or psychiatric disease; diabetes or other endocrine disease; immunosuppression
* Current treatment with medication or medical devices which affect GI motility and transit time (prokinetics, antidiarrheals, laxatives)
* Current treatment with medication which affect glucose metabolism or appetite
* Current treatment with beta blockers or peroral steroids
* Current treatment with non-steroidal anti-inflammatory drugs, tricyclic antidepressants, selective serotonin re-uptake inhibitors or opioids
* Bariatric surgery
* GI symptoms or diseases such as regular (weekly) abdominal pain, dysphagia, gastric bezoars, strictures, fistulas, bowel obstructions, diverticulitis, celiac disease, Crohn's disease, ulcerative colitis or proctitis
* Alcohol/drug abuse or in treatment with disulfiram (Antabus) at time of inclusion
* Pregnant or lactating women
* Fertile women not using birth control agents including oral contraceptives, gestagen injection, subdermal implants, hormonal vaginal ring, transdermal application, or intra-uterine devices
* Concomitant participation in other research studies

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time (minutes) | Within 24 hours from ingestion of the SmartPill™ at both visits (standard breakfast meal and SmartBar™, respectively)
  Measured by the SmartPill™ technique. The SmartPill™ is ingested at both visits in combination with the standard breakfast meal and SmartBar™, respectively. The time frame depends on the individual gastric emptying time.

SECONDARY OUTCOMES:
Small bowel transit time (minutes) | Within 5 days after both visits (standard breakfast meal and SmartBar™, respectively)
  Measured by the SmartPill™ technique. The SmartPill™ is ingested at both visits in combination with the standard breakfast meal and SmartBar™, respectively. The time frame depends on the individual transit time.
Large bowel transit time (minutes) | Within 5 days after both visits (standard breakfast meal and SmartBar™, respectively)
  Measured by the SmartPill™ technique. The SmartPill™ is ingested at both visits in combination with the standard breakfast meal and SmartBar™, respectively. The time frame depends on the individual transit time.
Total gastrointestinal transit time (minutes) | Within 5 days after both visits (standard breakfast meal and SmartBar™, respectively)
  Measured by the SmartPill™ technique. The SmartPill™ is ingested at both visits in combination with the standard breakfast meal and SmartBar™, respectively. The time frame depends on the individual transit time.
Motility index (arbitrary unit) | Within 5 days after both visits (standard breakfast meal and SmartBar™, respectively)
  Calculated based on amplitudes and number of contractions measured using the SmartPill™ technique. The greater the motility index the greater the gastrointestinal motility (i.e. more frequent and stronger contractions). A higher motility index has been observed among healthy participants compared to patients with diabetic gastroparesis indicating that a higher index is favorable.
Metabolites | 0 minutes (fasting) and 15, 30, 45, 60, 90, 120, 180, 240 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Concentrations of metabolites (including but not limited to: glucose, lipids, cholesterol, free-fatty acids, and amino acids. Measured at both visits in the fasting state and for 4 hours after consumption of the standard breakfast meal and the SmartBar™, respectively.
Hormones | 0 minutes (fasting) and 15, 30, 45, 60, 90, 120, 180, 240 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Concentrations of hormones related to regulation of appetite, glucose and lipid metabolism (including but not limited to: insulin, glucagon, ghrelin, glucagon-like peptide-1 (GLP-1), glucose-dependent insulinotropic polypeptide (GIP) and peptide YY (PYY), leptin, fibroblast growth factor 19 (FGF-19), fibroblast growth factor 21 (FGF-21), growth differentiation factor 15 (GDF-15)).
Attention measured using eye tracking | 0 minutes (fasting) at 60 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Eye tracking metrics including gaze duration bias, gaze direction bias, fixations, saccades, pupil size/dilation, distance to screen, ocular vergence and blinks to measure attention in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire
Arousal measured using galvanic skin response | 0 minutes (fasting) and after 60 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Changes in conductivity of skin (galvanic skin response) in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire
Emotions measured using facial expression analysis | 0 minutes (fasting) and after 60 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Facial expression analyses using computer-vision algorithms (AFFDEX) to measure emotions in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire
Food choice | 0 minutes (fasting) and after 60 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Food choice is determined based on frequency of selection made within each food category. The scores range from 0-48 i.e. 0 = foods within a specific food category have not been selected at all to 48 = foods within a specific food category have been selected 48 times.
Implicit wanting | 0 minutes (fasting) and after 60 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Implicit wanting of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Implicit wanting is assessed based on food choice and response time for selected and non-selected food items as well as mean response time.
Explicit liking | 0 minutes (fasting) and after 60 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Explicit liking of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Explicit liking is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how pleasant would it be to taste this food right now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Explicit wanting | 0 minutes (fasting) and after 60 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Explicit wanting of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Explicit wanting is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how much do you want some of this food now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Subjective appetite | 0 minutes (fasting) and 15, 30, 45, 60, 90, 120, 180, 240 minutes (after consumption of the standard breakfast meal and SmartBar™, respectively)
  Rated using visual analogue scales and includes sensations of: Hunger, fullness, satiety, prospective food consumption, wellbeing, nausea, thirst, desire to eat meat, salty, and sweet. The scale range is 0-100 and each end represent the extremes e.g. hunger rating: "I am not hungry at all" to "I have never been this hungry before".
Self-reported gastrointestinal symptoms (part 1) | Answered during test days (0-240 minutes)
  Assessed from the questionnaire the Gastrointestinal Symptom Rating Scale (GSRS). Rated on 7-point likert scales. Range: 1 = absence of symptoms to 7 = very severe symptoms.
Self-reported gastrointestinal symptoms (part 2) | Answered during test days (0-240 minutes)
  Assessed from the Gastrointestinal Symptom Score (PAGI-SYM). Rated on 6-point likert scales. Range: 1 = absence of symptoms to 6 = very severe symptoms.
Self-reported gastrointestinal symptoms (part 3) | Registered 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Number of symptoms. Assessed from logs.
Self-reported autonomic symptoms | Answered during test days (0-240 minutes)
  Assessed from the questionnaire COMPASS31
Body weight (kg) | At 0 minutes (fasting) at both visits
  Body weight is measured on a digital scale
Body mass index (kg/m^2) | At 0 minutes (fasting) at both visits
  Calculated from body weight (kg) and height (m)
Fat mass (kg) | At 0 minutes (fasting) at both visits
  Measured by Dual-energy X-ray Absorptiometry
Fat percentage (%) | At 0 minutes (fasting) at both visits
  Measured by Dual-energy X-ray Absorptiometry
Fat free mass (kg) | At 0 minutes (fasting) at both visits
  Measured by Dual-energy X-ray Absorptiometry
Waist circumference (cm) | At 0 minutes (fasting) at both visits
  Measured using tape measure
Hip circumference (cm) | At 0 minutes (fasting) at both visits
  Measured using tape measure
Mean amplitude of glycaemic excursions (MAGE) | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Measured using continous glucose monitoring
Continuous overall net glycaemic action (CONGA) | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Measured using continous glucose monitoring
Daily time spent above different glucose concentrations (e.g. >6.1 mmol/L, >7.0 mmol/L, >7.8 mmol/L, and >11.1 mmol/L) | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Measured using continous glucose monitoring
Mean glucose concentrations | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Measured using continous glucose monitoring
Standard deviation of glucose concentrations | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Measured using continous glucose monitoring
Variation coefficients of glucose concentrations | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Measured using continous glucose monitoring
Resting energy expenditure (kcal/day) | At 0 minutes (fasting) at both visits
  Measured by indirect calorimetry under resting and fasting conditions
Substrate oxidation (respiratory exchange ratio) | At 0 minutes (fasting) at both visits
  Measured by indirect calorimetry under resting and fasting conditions
Systolic blood pressure (mmHg) | At 0 minutes (fasting) at both visits
  Measured under resting and fasting conditions
Diastolic blood pressure (mmHg) | At 0 minutes (fasting) at both visits
  Measured under resting and fasting conditions
Heart rate (bpm) | At 0 minutes (fasting) at both visits
  Measured under resting and fasting conditions during measurements of blood pressure and in the supine position by a handheld ECG measuring device (Vagus™).
Heart rate response to standing up from the supine position | At 0 minutes (fasting) at both visits
  Measured by a handheld ECG measuring device (Vagus™).
Heart rate response to inhalation and exhalation | At 0 minutes (fasting) at both visits
  Measured by a handheld ECG measuring device (Vagus™).
Heart rate response to forced exhalation during rest (valsalva maneuver) | At 0 minutes (fasting) at both visits
  Measured by a handheld ECG measuring device (Vagus™).
Microbiome content and diversity | One sample during 6 days after both visits
  Determined from stool samples. Bacterial DNA and RNA will be purified from the stool samples and changes in the microbiome composition and function will be estimated based on sequencing of the microbiomes' DNA and RNA. Includes but is not limited to the Firmicutes/Bacteroidetes ratio.
Physical activity (time spent at different intensities) | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Sedentary time, light, moderate and vigorous intensity physical activity. Assessed from 24 h/day accelerometry
Physical activity (counts/min) | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from 24 h/day accelerometry
Physical activity energy expenditure (kcal/day) | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from 24 h/day accelerometry
Physical activity (MET hours) | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from 24 h/day accelerometry
Timing of physical activity (hh:mm) | Measured for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from activity logs and 24 h/day accelerometry
Energy intake (kcal/day) | Assessed for 3 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from diet records
Macronutrient intake (energy percentage) | Assessed for 3 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from diet records
Timing of dietary intake (hh:mm) | Assessed for 3 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from diet records
Sleep timing (hh:mm) | Assessed for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Including bedtime, sleep onset, wake-up, time out of bed, sleep midpoint. Assessed from sleep logs and 24 h/day accelerometry
Sleep duration (minutes) | Assessed for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from sleep logs and 24 h/day accelerometry
Sleep variability (minutes) | Assessed for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Variability in bedtime, wake-up, sleep duration and sleep midpoint. Assessed from sleep logs and 24 h/day accelerometry
Sleep onset latency (minutes) | Assessed for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from sleep logs and 24 h/day accelerometry
Sleep efficiency (%) | Assessed for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from 24 h/day accelerometry
Wakefulness (minutes) | Assessed for 6 days after both visits (standard breakfast meal and the SmartBar™ conditions)
  Assessed from 24 h/day accelerometry
HbA1c (mmol/mol and %) | At 0 minutes at both visits
  Hemoglobin A1c
Insulin sensitivity (indices) | At 0 minutes (fasting) and 4 hours after consumption of the standard breakfast meal and the SmartBar™, respectively
  Including but not limited to the Matsuda index
Insulin resistance (indices) | At 0 minutes (fasting) and 4 hours after consumption of the standard breakfast meal and the SmartBar™, respectively
  Including but not limited to Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Færch, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Jensen MM, Pedersen HE, Clemmensen KKB, Ekblond TS, Ried-Larsen M, Faerch K, Brock C, Quist JS. Associations Between Physical Activity and Gastrointestinal Transit Times in People with Normal Weight, Overweight, and Obesity. J Nutr. 2024 Jan;154(1):41-48. doi: 10.1016/j.tjnut.2023.06.005. Epub 2023 Jun 12. PMID 37315794